CLINICAL TRIAL: NCT06769529
Title: Observational Cohort Study of Adult Patients With Congenital Heart Disease
Acronym: ACHD-BO
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ACHD-BO
Record Dates: First submitted 2024-11-28; First posted 2025-01-10 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-11

CONDITIONS: Adult Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 11 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this retrospective and prospective single-center observational study is to evaluate the correct management of adult patients with congenital heart diseas (ACHD), based on the experience of a reference center such as the Institute of Pediatric Cardiology at Policlinico Sant'Orsola Malpighi. The patients participating in this study will not be subjected to any procedures beyond normal daily clinical practice; likewise, the clinical variables that will be collected for the study are those that are commonly collected by the physician in daily clinical practice. This study therefore involves naturalistic observation of current clinical practice without the application of any kind of intervention.

DETAILED DESCRIPTION:
To date, there are an estimated 1 million patients, a population that is expected to grow by about 5%.annually. Given the increase in the number of such patients and their complexity, there is an increasing need to train experienced cardiologists and cardiac surgeons.

Our study is part of this panorama with the aim of assessing the correct management, taking into account the important psychological and sociological impact of these diseases, based on the experience of a reference centre such as the Institute of Paediatric Cardiology of the Policlinico Sant'Orsola Malpighi. The primary objective of the study is to identify the clinical and epidemiological characteristics of adult patients with heart disease congenital heart disease (in natural history or previously undergoing corrective or palliative intervention) and to define the need for intervention at a distance, both in terms of interventional and surgical procedures. 1) to describe cardiovascular adverse events and mortality in the target population during follow-up and any non-cardiac comorbidities; 2) to provide data defining the level of utilisation of healthcare resources (diagnostic tests withhigh complexity/cost diagnostic tests, hospital admissions, hospital admissions in high intensity wardscare, percutaneous interventional procedures, surgical procedures); 3) to assess data on quality of life, reproductive health (for the sub-population of female sub-population).

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital heart disease in natural history or previously undergoing palliative or corrective surgery in the time period after 14/02/2014
* Obtaining informed consent

Exclusion Criteria:

* Age < 18 years
* Inability to obtain longitudinal data after the first follow-up performed at our Center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study includes all patients with congenital heart disease and age older than 18 years, referred to our Pediatric Cardiology Center from 14 February 2014 to 01 May 2025 going to represent one for a cohort of about 2000 patients.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Patient's medical history and diagnosis | Through study duration, an average of 10 years
  Anthropometric data (age, sex, weight, height, body surface area) Detailed cardiologic diagnosis classified according to anatomic complexity Presence of univentricular physiology The presence of a genetic syndrome, or reasonable suspicion of its presence Major comorbidities The surgical and interventional cardiology history The level of urgency of admission to the department and the hemodynamics room Pregnancies prior to the visit The physiologic status Sinus rhythm Therapy
Clinical events | Through study duration, an average of 10 years
  History of syncope since first evaluation History of NYHA III/IV since first evaluation History of moderate-grade left ventricular dysfunction History of severe grade left ventricular dysfunction Cyanosis History of cerebrovascular events (stroke/transient ischemic attack) History of endocarditis History of ventricular arrhythmias that required medical intervention History of supraventricular arrhythmias that required medical intervention Pace-Maker Implantation Implantation of Defibrillator (ICD) Implantation of Defibrillator-Resynchronizer (ICD-CRT)
Patient visits, diagnostic tests, hospitalizations, and interventions | Through study duration, an average of 10 years
  Longitudinal clinical evaluations Longitudinal advanced imaging assessments Longitudinal hospitalizations oIndications for hospitalization Longitudinal transcatheter procedures Type of transcatheter procedure Longitudinal surgical procedures Type of surgical procedure
Clinical events after cardiology evaluation | Through study duration, an average of 10 years
  Death Ventricular arrhythmia with need for intervention Supraventricular arrhythmia with need for intervention Progression to NYHA functional class III/IV Unscheduled hospitalization Bleeding Development of pulmonary hypertension Cerebrovascular event (stroke/transient ischemic attack) Plastic bronchitis Protido-dispersing enteropathy Failure of Fontan circulation Evaluation for cardiac transplantation
  * Refusal for cardiac transplantation
  * Listing for cardiac transplantation
  * Endocarditis
  * Cardiac transplantation
The manner of death | Through study duration, an average of 10 years
  Sudden cardiac death Heart death from heart failure Cardiac death related to surgical procedure Cardiac death related to transcatheter procedure Cardiac death from cerebrovascular event Cardiac death from endocarditis or sepsis Noncardiac neoplastic Noncardiac by renal failure Noncardiac by suicide Other noncardiac modality

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Egidy Assenza, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy